CLINICAL TRIAL: NCT00954811
Title: A Phase IV Study on the Effect of Luteal Supplementation With Rec-LH on the Pregnancy Rate After Ovulation Triggering With GnRH-agonist Instead of HCG in IVF Protocol;Proof of Concept
Brief Title: Luteal Supplementation With Rec-LH After GnRH-agonist Triggering in In Vitro (IVF)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Dr Papanikolaou Evangelos, Centre for Reproductive Medicine,UZ Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: recombinant LH 1505
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2009-08

CONDITIONS: Pregnancy; Pregnancy Loss
Keywords: pregnancy
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HCG for ovulation triggering and luteal progesterone (Active Comparator): conventional triggering with HCG and conventional luteal support with progesterone
  Interventions: Drug: progesterone 600mg
- Agonist triggering and rec-LH luteal support plus progesterone (Experimental): new method of triggering with GnRH-agonist and proof of concept intervention with novel way of luteal support with rec-LH plus the usual co-treatment with progesterone
  Interventions: Drug: 300IU rec-LH

INTERVENTIONS:
Drug: 300IU rec-LH — luteal alternate doses
  Arms: Agonist triggering and rec-LH luteal support plus progesterone
Drug: progesterone 600mg — luteal support
  Arms: HCG for ovulation triggering and luteal progesterone

SUMMARY:
Our aim is to access whether we can achieve equivalent pregnancy rates by the addition of six doses of luteal support with recLH after agonist triggering for IVF cycles in the absence of OHSS.

DETAILED DESCRIPTION:
Whether pregnancy outcome after GnRH-agonist triggering could be improved by adding luteal recLH support plus progesterone, compared to that observed after ovulation triggering with HCG in GnRH antagonist stimulated cycles.

ELIGIBILITY:
Inclusion Criteria:

* < 36years,
* single blastocystET,
* FSH < 12

Exclusion Criteria:

* endometriosis,
* 3 and 4,
* pco,
* frozen sperm

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-01 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
pregnancy occurrence, pregnancy loss | 14 days after OPU

SECONDARY OUTCOMES:
hormone levels, OHSS, endometrium | 14 days after oocyte pick up

CONTACTS AND LOCATIONS:
Overall Officials: Paul Devroey, Study Chair — Professor or OB-GYN
Locations (1):
- Centre for Reproductive Medicine, UZ Brussel, Brussels, Jette, Belgium